CLINICAL TRIAL: NCT07355153
Title: Feasibility and Preliminary Effectiveness of 'Managing Cancer and Living Meaningfully'
Brief Title: Feasibility of CALM Therapy in Korean Cancer Patients
Acronym: CALM_Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Kyungpook National University Chilgok Hospital (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jungmin Woo, Professor, Kyungpook National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNUH 2019-05-028; KNUCH 2019-04-026-001 (Other: Kyungpook National University Chilgok Hospital)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Depression
Keywords: Quality of life; Depression; Cancer; Psychotherapy; Behavioral symptoms
MeSH Terms: conditions — Depression; Neoplasms; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility study with mixed-methods evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CALM Therapy (Experimental): Participants receive 3-6 individual CALM therapy sessions over 3-6 months
  Interventions: Behavioral: Managing Cancer and Living Meaningfully (CALM)

INTERVENTIONS:
Behavioral: Managing Cancer and Living Meaningfully (CALM) — CALM (Managing Cancer and Living Meaningfully) is a semi-structured, manualized individual psychotherapy designed for patients with advanced cancer, grounded in relational, attachment, and existential theory.
  CALM consists of 3-6 individual sessions (45-60 minutes each) delivered over 3-6 months by specially trained therapists. The therapy addresses four core domains: (1) symptom management and communication with healthcare providers; (2) changes in self and relations with close others; (3) sense of meaning and purpose; and (4) the future and mortality. All domains are addressed with each patient, with sequencing and emphasis tailored to individual concerns.
  Patients' caregivers or family members are encouraged to participate in sessions as appropriate. CALM can be delivered by trained therapists from various disciplines including psychiatry, psychology, social work, nursing, and medicine.

SUMMARY:
This feasibility study examined the cultural adaptation and implementation of Managing Cancer and Living Meaningfully (CALM) therapy for advanced cancer patients in Korea. CALM is a brief manualized individual psychotherapy designed to address psychological distress and existential concerns in patients with advanced disease.

DETAILED DESCRIPTION:
This single-arm feasibility study evaluated the acceptability, tolerability, and preliminary effectiveness of CALM therapy in the Korean cultural and healthcare context. Patients with advanced or metastatic solid-tumor cancers received 3-6 individual therapy sessions over 3-6 months, delivered by trained psychiatrists.

The study assessed feasibility through recruitment rates, therapy completion rates, and outcome measure completion. A mixed-methods approach included quantitative outcome measures (depression, death anxiety, attachment, quality of life, anxiety) and qualitative interviews with patients and caregivers to evaluate implementation barriers and facilitators.

This study was conducted in collaboration with the developers of CALM therapy at Princess Margaret Cancer Centre, Toronto, Canada. Therapists were trained through the international CALM training program, including workshop attendance and supervised training cases under the supervision of the intervention developers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* Fluent in Korean
* Able to provide informed consent
* Diagnosis of advanced or metastatic solid-tumor cancer, including:

  * Stage III or IV lung or ovarian cancer
  * Any stage of pancreatic cancer
  * Stage IV gastrointestinal, gynecological, breast, genitourinary, sarcoma, melanoma, or endocrine cancer
  * Unresectable cholangiocarcinoma, liver, ampullary, or peri-ampullary cancer

Exclusion Criteria:

* Major communication difficulties
* Inability to commit to 3-6 psychotherapy sessions (e.g., too ill to participate, lack of transportation, insufficient motivation)
* Cognitive impairment as indicated by clinical team or patient chart

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rate | 2 years (June 2019 - June 2021)
  Recruitment of at least 51 patients over 2 years
Feasibility: Outcome Measure Completion Rate | Through study completion, up to 6 months per participant
  At least 66% of patients complete the outcome measures at least 50% of the time
Feasibility: Therapy Completion Rate | Through study completion, up to 6 months per participant
  At least 50% of patients complete at least 3 CALM sessions

SECONDARY OUTCOMES:
Depression Symptoms (PHQ-9) | Baseline, 3 months, and 6 months
  Patient Health Questionnaire-9, a 9-item measure of depression. Scores range 0-27, with higher scores indicating more severe depressive symptoms.
Death-Related Distress (DADDS) | Baseline, 3 months, and 6 months
  Death and Dying Distress Scale, a validated 15-item scale measuring death anxiety in advanced cancer patients, addressing fears about the dying process and distress about lost opportunities and self-perceived burden.
Attachment Security (ECR-M16) | Baseline, 3 months, and 6 months
  Modified and brief Experiences in Close Relationships scale, a 16-item measure of attachment security assessing attachment anxiety (fear of abandonment) and avoidance (defensive independence). Lower scores indicate greater attachment security.
Quality of Life (QUAL-EC) | Baseline, 3 months, and 6 months
  Quality of Life at the End of Life-Cancer Scale, measuring quality of life in patients near end of life. Includes 4 subscales: Symptom Impact, Preparation for End-of-Life, Relationship with Healthcare Providers, and Life Completion.
Treatment Evaluation (CEQ) | 3 months and 6 months
  Modified Clinical Evaluation Questionnaire, a 15-item measure (7 original + 8 added items) evaluating the extent to which patients felt supported by their CALM therapist and how CALM therapy helps patients cope with the future, discuss important things with loved ones, and increase double awareness.
Generalized Anxiety (GAD-7) | Baseline, 3 months, and 6 months
  Generalized Anxiety Disorder-7, a 7-item measure of anxiety symptoms. Scores range 0-21, with higher scores indicating more severe anxiety.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Rodin G, Lo C, Rydall A, Shnall J, Malfitano C, Chiu A, Panday T, Watt S, An E, Nissim R, Li M, Zimmermann C, Hales S. Managing Cancer and Living Meaningfully (CALM): A Randomized Controlled Trial of a Psychological Intervention for Patients With Advanced Cancer. J Clin Oncol. 2018 Aug 10;36(23):2422-2432. doi: 10.1200/JCO.2017.77.1097. Epub 2018 Jun 29. PMID 29958037